CLINICAL TRIAL: NCT00021918
Title: Serum Total Homocysteine and C-Reactive Protein - Ancillary to IDNT
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 975; R01HL067695 (NIH)
Record Dates: First submitted 2001-08-10; First posted 2001-08-10 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-10

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Heart Diseases; Diabetes Mellitus, Non-insulin Dependent; Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Heart Diseases; Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To examine the independent association of serum total homocysteine and C-reactive protein with arteriosclerotic cardiovascular disease morbidity and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Patients with diabetic nephropathy experience markedly increased rates of morbidity and mortality due to arteriosclerotic cardiovascular disease [CVD]. Established arteriosclerotic risk factors such as age, sex, cigarette smoking, hypertension, and dyslipidemia do not account adequately for this excess CVD risk. Prospective data from general populations, and much more limited findings from both diabetic cohorts. and cohorts with chronic renal disease, have linked elevated levels of total homocysteine (tHcy) and C-reactive protein (CRP) to arteriosclerotic CVD morbidity and mortality. Determination of baseline serum total homocysteine and C-reactive protein concentrations in the Irbesartan Type 2 Diabetic Nephropathy Trial (IDNT) cohort affords a truly unique opportunity to evaluate the potential independent relationship between these putative CVD risk factors and subsequent CVD morbidity and mortality, in this patient population. The IDNT is a multicenter, randomized, double-blind, placebo-controlled trial of 1,715 hypertensive, Type 2 diabetic patients aged 30 to 70 who have overt nephropathy (24 hour urinary protein excretion greater than 900 mg and a serum creatinine of 90 to 265 micromols/L). The IDNT compares the effect of the angiotensin II receptor antagonist irbesartan with placebo and amlodipine on the progression of renal disease and mortality. The IDNT is supported by Bristol-Myers Squibb Company in Princeton, New Jersey and Sanofi-Synthelabo in Paris, France.

The study is in response to an initiative "Ancillary Studies in Heart, Lung, and Blood Disease Trials" released by the National Heart, Lung, and Blood Institute in June 2000.

DESIGN NARRATIVE:

The first specific aim is to conduct longitudinal analyses of the potential "Independent" relationship between baseline concentrations of serum total homocysteine and C-reactive protein in the full IDNT cohort, and subsequent:pooled cardiovascular disease morbidity and mortality (primary analysis). total mortality, (after multivariable -adjustment for the established predictors of cardiovascular disease morbidity/ mortality, and total mortality). The second specific aim is to conduct cross-sectional analyses to assess baseline serum total homocysteine and C-reactive protein concentrations in the full IDNT cohort, in relation to potential baseline determinants of these analytes, including: B-vitamin status; age and gender; renal function indices, i.e. both creatinine-based glomerular filtration rate estimates, and proteinuria; indices of glycemia, prevalent cardiovascular disease (CVD), traditional CVD risk factors (i.e., in particular, smoking, blood pressure, and total cholesterol/HDL cholesterol ratio).

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bostom — Memorial hospital

REFERENCES:
- [Background] Friedman AN, Hunsicker LG, Selhub J, Bostom AG. Clinical and nutritional correlates of C-reactive protein in type 2 diabetic nephropathy. Atherosclerosis. 2004 Jan;172(1):121-5. doi: 10.1016/j.atherosclerosis.2003.09.011. PMID 14709365
- [Background] Friedman AN, Hunsicker LG, Selhub J, Bostom AG; Collaborative Study Group. Total plasma homocysteine and arteriosclerotic outcomes in type 2 diabetes with nephropathy. J Am Soc Nephrol. 2005 Nov;16(11):3397-402. doi: 10.1681/ASN.2004100846. Epub 2005 Sep 14. PMID 16162814
- [Background] Friedman AN, Hunsicker LG, Selhub J, Bostom AG; Collaborative Study Group. C-reactive protein as a predictor of total arteriosclerotic outcomes in type 2 diabetic nephropathy. Kidney Int. 2005 Aug;68(2):773-8. doi: 10.1111/j.1523-1755.2005.00456.x. PMID 16014055